CLINICAL TRIAL: NCT06722014
Title: Integrating Pain-CBT Into an mHealth Analgesic Support Intervention for Patients With Chronic Pain From Advanced Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Desiree R. Azizoddin PsyD, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-286; 5K08CA266937 (NIH)
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Pain; Pain Syndrome; Advanced Cancer
Keywords: Pain; Pain Syndrome; Advanced Cancer
MeSH Terms: conditions — Pain; Somatoform Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort C: STAMP + CBT App (Experimental): Permutated-block randomization and a block size of 6 will be used to randomize 60 participants to this cohort, and participants will complete:
  * Baseline in-person or remote visit with an introduction to the STAMP+CBT application.
  * Surveys via the application 6 days per week.
  * Day 7 check in with study team
  * Day 14 survey
  * Day 28 follow-up surveys
  * Optional in-person or remote semi-structured, exit interview
  * Day 42 (Week 6) follow-up survey
  Interventions: Behavioral: STAMP + CBT
- Cohort D: Digital Cancer Pain Education Packet + Usual Care (Other): Permutated-block randomization and a block size of 6 will be used to randomize 60 participants to this cohort, and participants will complete:
  * Baseline in-person or remote visit with introduction to the digital cancer pain education packet and pain tracker form.
  * Completion of pain tracker
  * Day 7 check in with study team
  * Day 14 survey
  * Day 28 surveys
  * Optional in-person or remote semi-structured, exit interview to review the educational packet
  * Day 42 (Week 6) follow-up survey
  Interventions: Behavioral: Digital Cancer Pain Education Packet

INTERVENTIONS:
Behavioral: STAMP + CBT — A mobile health, smartphone application that provides tailored multi-media, cancer pain psycho-education and pain management coping skills using algorithm-based technology to provide in the moment symptom monitoring and feedback.
  Other Names: Smartphone Technology to Alleviate Malignant Pain+Cognitive Behavioral Therapy for pain
  Arms: Cohort C: STAMP + CBT App
Behavioral: Digital Cancer Pain Education Packet — Packet including Articles from the Association for Clinical Oncology and the National Cancer Institute and the pain and medication monitoring form.
  Arms: Cohort D: Digital Cancer Pain Education Packet + Usual Care

SUMMARY:
Smartphone Technology to Alleviate Malignant Pain (STAMP) + Cognitive Behavioral Therapy for Pain (STAMP+CBT) The purpose of the study is to develop and refine the mHealth pain-CBT app intervention and carry out a randomized pilot to test the novel mHealth (Mobile health technology) intervention, which harmonizes psychological and pharmacological support for advanced cancer pain.

The name of the study smartphone application involved in this study is:

-STAMP+CBT

DETAILED DESCRIPTION:
The purpose of the study is to make sure the app is usable and helpful for participants with cancer and to get feedback about participants experiences after using the app for four weeks. Outcomes related to pain, quality of life, and healthcare utilization will also be assessed. The cancer pain education packet and pain and medication monitoring survey are standard care. The app is intended to improve self-management of cancer-related pain.

The study will begin with Cohort A, followed by Cohort B. These two cohorts are to refine the STAMP+CBT intervention. Then a randomized pilot will be performed, and participants will be randomized into one of two study groups for the pilot: Cohort C: STAMP+CBT versus Cohort D: Digital Cancer Pain Education Packet + Usual Care. Randomization means a participant is placed into a study group by chance.

It is expected that about 60 people will take part in this research study.

The National Institutes of Health, National Cancer Institute (NIH-NCI), is funding this research study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 years
* Patient diagnosed with an active cancer diagnosis (locally advanced solid tumor malignancy, multiple myeloma, or other advanced hematologic malignancy), either undergoing active treatment or receiving treatment for an advanced cancer or are receiving supportive/palliative care
* Chronic pain related to cancer or treatment (> pain score of 4 on a 0-10 scale)
* Has an active prescription for at least one opioid medication to treat their cancer pain (i.e. not for post-surgical pain)
* Own/use a compatible smartphone (iPhone or Android)

Exclusion Criteria:

* Patients in survivorship: patients who have completed their treatment regimens, are not actively receiving treatment for an advanced cancer, or have a cancer that is in remission
* Cognitive impairment that would interfere with study participation, as judged by treating clinician (e.g. delirium, dementia)
* Inability to speak English (the intervention has not yet been translated to Spanish)
* Currently in CBT treatment
* Enrolled in hospice
* Currently hospitalized
* Use of transmucosal fentanyl, given safety concerns and ongoing risk mitigation program required to prescribe these (TIRF REMS)
* Pain primarily related to a recent surgery (within the last 2 weeks)
* Conditions that hinder smartphone use
* The study will exclude adults who are unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, and prisoners.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall intervention adherence rate (Cohort C) | Up to 4 weeks
  >70% of subjects complete any activity on the STAMP+CBT application at least 50% of days on study (4-week study period). The app will be considered feasible if this benchmark is achieved.
Overall intervention adherence rate (Cohort D) | Up to 4 weeks
  Defined as completion of the 14- and 28-days surveys, which assesses completion of the pain and medication monitoring reports by participants in the control group.
Proportion of participants who rate app acceptability at least 4/5 on the Acceptability E-Scale (Cohort C) | Up to 6 weeks
  Acceptability of the intervention is defined as > 80% of the participants rate the application as satisfactory and useful with a mean 4 or higher score out of 5 on the Acceptability E-Scale (Tariman 2011). The Acceptability E-Scale a 7-item measure with answer ranging from 1 "Very Difficulty/Difficult to understand/Not at all/Very unacceptable/Very dissatisfied/Not useful/Very unlikely" to 5 "Very Easy/Easy to understand/Very much/ Very acceptable/Very satisfied/Very useful/Very likely" and with a total scores range of 7 to 35 with a higher score representing greater participant acceptability. Subjects will be assigned surveys at baseline, 4 weeks, and 6 weeks. Participants will rate the app on the following 5 domains: understandability, enjoyability, ease of use, time required to use the app, and overall satisfaction. Ratings lower than 4/5 will lead to refinements.
Proportion of participants who rate educational packet acceptability at least 4/5 on the Acceptability E-Scale (Cohort D) | Up to 6 weeks
  Acceptability of the intervention is defined as > 80% of the participants rate the application as satisfactory and useful with a mean 4 or higher score out of 5 on the Acceptability E-Scale (Tariman 2011). The Acceptability E-Scale a 7-item measure with answer ranging from 1 "Very Difficulty/Difficult to understand/Not at all/Very unacceptable/Very dissatisfied/Not useful/Very unlikely" to 5 "Very Easy/Easy to understand/Very much/ Very acceptable/Very satisfied/Very useful/Very likely" and with a total scores range of 7 to 35 with a higher score representing greater participant acceptability. Subjects will be assigned surveys at baseline, 4 weeks, and 6 weeks. Participants will rate the app on the following 5 domains: understandability, enjoyability, ease of use, time required to use the app, and overall satisfaction. Ratings lower than 4/5 will lead to refinements.

SECONDARY OUTCOMES:
Number of Enrolled Participants who Consented and Completed the Study (Cohort C) | 18 months
  Defined as the proportion of participants of the intervention group on study for the complete study period. Subjects are defined as individuals who consented and enrolled to the trial and complete study measures and either 28 days of app use (intervention group) or 28 days of education packet review (control group). Rates of completion will be compared between the intervention and control groups.
Number of Enrolled Participants who Consented and Completed the Study (Cohort D) | 18 months
  Defined as the proportion of participants of the control group on study for the complete study period. Subjects are defined as individuals who consented and enrolled to the trial and complete study measures and either 28 days of app use (intervention group) or 28 days of education packet review (control group). Rates of completion will be compared between the intervention and control groups.
Study Retention (Cohort C) | 18 months
  Defined as the proportion of participants of the intervention group on study for the complete study period. Subjects are defined as individuals who consented and enrolled to the trial and complete study measures and either 28 days of app use (intervention group) or 28 days of education packet review (control group). Rates of completion will be compared between the intervention and control groups.
Study Retention (Cohort D) | 18 months
  Defined as the proportion of participants of the control group on study for the complete study period. Subjects are defined as individuals who consented and enrolled to the trial and complete study measures and either 28 days of app use (intervention group) or 28 days of education packet review (control group). Rates of completion will be compared between the intervention and control groups.
Median assessment score on the system usability scale at 4 weeks (Cohort C) | Up to 6 weeks
  Intervention usability will be assessed by the System Usability Scale (SUS), a 12-item measure rated on a 5-point Likert scale from 1 "Strongly Disagree" to 5 "Strongly Agree" with a total scores range of 0 to 100. A higher score represents greater usability. Subjects will be assigned surveys at baseline, 4 weeks, and 6 weeks. The survey at 4 weeks will assess intervention acceptability with the System Usability Scale (Brooke, 2002). The app will be considered usable if the median score on the System Usability Scale across respondents is >75.
Median assessment score on the system usability scale at 4 weeks (Cohort D) | Up to 6 weeks
  Intervention usability will be assessed by the System Usability Scale (SUS), a 12-item measure rated on a 5-point Likert scale from 1 "Strongly Disagree" to 5 "Strongly Agree" with a total scores range of 0 to 100. A higher score represents greater usability. Subjects will be assigned surveys at baseline, 4 weeks, and 6 weeks. The survey at 4 weeks will assess control education packet acceptability with the System Usability Scale (Brooke, 2002). This information will be used to compare usability scores across intervention and control groups.
Change in Brief Pain Inventory (BPI) Pain Interference Score from Baseline to 4 and 6 Weeks (Cohort C) | Up to 6 weeks
  Assessed by the BPI, a 7-item subscale on pain interference with answers scored on a scale from 0 "Does not interfere" to 10 "Greatly interferes." A total scores range is 0 to 70 with a higher score indicating greater pain interference.
Change in BPI Pain Interference Score from Baseline to 4 and 6 Weeks (Cohort D) | Up to 6 weeks
  Assessed by the BPI, a 7-item subscale on pain interference with answers scored on a scale from 0 "Does not interfere" to 10 "Greatly interferes." A total scores range is 0 to 70 with a higher score indicating greater pain interference.
Change in BPI Pain Intensity Score from Baseline to 4 and 6 Weeks (Cohort C) | Up to 6 weeks
  Assessed by the Brief Pain Inventory (BPI) pain intensity subscale, a 4-item measure on pain intensity with answers scored on a scale from 0 "No pain" to 10 "Pain as bad as you can imagine." A total scores range is 0 to 40 with a higher score indicating greater pain intensity.
Change in BPI Pain Intensity Score from Baseline to 4 and 6 Weeks (Cohort D) | Up to 6 weeks
  Assessed by the Brief Pain Inventory (BPI) pain intensity subscale, a 4-item measure on pain intensity with answers scored on a scale from 0 "No pain" to 10 "Pain as bad as you can imagine." A total scores range is 0 to 40 with a higher score indicating greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Desiree Azizoddine, PsyD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu